CLINICAL TRIAL: NCT03627455
Title: A Sex-specific Analysis of the Predictive Value of Troponin I and T in Patients With and Without Diabetes Mellitus After Successful Coronary Intervention
Brief Title: Troponin I and T and Adverse Outcomes in Patients With and Without Diabetes Mellitus After Coronary Intervention
Status: Completed | Type: Observational
Sponsor: Wilhelminenspital Vienna (Other)
Collaborators: Association for the Promotion of Research in Atherosclerosis, Thrombosis and Vascular Biology (Other)
Responsible Party: Principal Investigator, Maximilian Tscharre, MD, Principal Investigator, Wilhelminenspital Vienna
Other Study IDs: TROPDM2GENDER
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Male, with DM
  Interventions: Other: Percutaneous coronary intervention
- Male, without DM
  Interventions: Other: Percutaneous coronary intervention
- Female, with DM
  Interventions: Other: Percutaneous coronary intervention
- Female, without DM
  Interventions: Other: Percutaneous coronary intervention

INTERVENTIONS:
Other: Percutaneous coronary intervention — Percutaneous coronary intervention

SUMMARY:
Elevated levels of troponin are associated with future MACE. Data on the prognostic value of high sensitive troponin T (hs-TnT) as compared to high sensitive troponin I (hs-TnI) in diabetic and non-diabetic patients are sparse.

We aimed to assess the risk for MACE according to gender and diabetes status and to compare the prognostic value of hs-TnT and hs-TnI with regards to clinical outcomes in diabetic and non-diabetic patients undergoing percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Percutaneous coronary intervention

Exclusion Criteria:

* unsuccessful percutaneous coronary intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients undergoing percutaneous coronary intervention at the department of cardiology at the Wihelminenspital
Sampling Method: Non-Probability Sample
Enrollment: 818 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
MACE | 8 years
  All-cause death, non-fatal myocardial infarction, non-fatal stroke

IPD SHARING:
Plan to Share IPD: Undecided